CLINICAL TRIAL: NCT00943267
Title: Effect of Intrapulmonary Administration of Recombinant Human Activated Protein C on Local Coagulation and Inflammation After Bronchial Instillation of Lipopolysaccharide in Humans
Brief Title: Effect of Intrapulmonary Recombinant Human Activated Protein C (APC) on Coagulation and Inflammation After Lipopolysaccharide (LPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Tom van der Poll MD PhD, Center for Experimental Molecular Medicine, AMC-UvA, Amsterdam, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CEMM-APC-01; MEC 08/188
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2009-07

CONDITIONS: Pneumonia; Lipopolysaccharides
Keywords: Activated Protein C; Lipopolysaccharides; Inflammation, Pulmonary
MeSH Terms: conditions — Pneumonia | interventions — Sodium Chloride; Endotoxins; Bronchoscopy; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activated protein C (Experimental)
  Interventions: Drug: Drotrecogin alpha; Drug: Endotoxin; Procedure: Bronchoscopy; Procedure: Blood sampling
- Saline (Placebo Comparator)
  Interventions: Drug: Saline (NaCl 0.9%); Drug: Endotoxin; Procedure: Bronchoscopy; Procedure: Blood sampling

INTERVENTIONS:
Drug: Drotrecogin alpha — Drotrecogin alpha is given intrabronchially by bronchoscopy at t=0
  Arms: Activated protein C
Drug: Saline (NaCl 0.9%) — Normal saline is given intrabronchially by bronchoscopy at t=0
  Arms: Saline
Drug: Endotoxin — Endotoxin (4 ng/kg body weight) is given intrabronchially in one subsegment at t=0
Procedure: Bronchoscopy — Bronchoscopies are performed at t=0 (for instillation of LPS and Drotrecogin alpha) and at t=6 (for performing a bronchoalveolar lavage)
Procedure: Blood sampling — Blood sampling is done by venapuncture at t=0 and t=6

SUMMARY:
Recombinant human Activated Protein C (rhAPC) has been shown to reduce the mortality of patients with severe sepsis. The biological effects of APC are pleiotropic, and can be roughly divided in anticoagulant and cytoprotective effects. Lung infection and inflammation are associated with reduced bronchoalveolar levels of endogenous APC. Recent evidence derived from animal studies indicates that local administration of rAPC into the lungs exerts local anti-inflammatory and anticoagulant effects. In this study we propose to study the potential of locally administered APC, within a lung subsegment, to inhibit lipopolysaccharide (LPS) induced lung inflammation and coagulation in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-35 years of age
* No clinically significant findings during physical examination and hematological and biochemical screening
* Normal spirometry and ECG
* Able to communicate well with the investigator and to comply with the requirements of the study
* No medication
* Written informed consent
* No smoking

Exclusion criteria:

* Known diseases
* A history of smoking within the last six months, or regular consumption of greater than three units of alcohol per day
* Administration of any investigational drug within 30 days of study initiation
* Donation of blood within 60 days, or loss of greater than 400 ml of blood within 12 weeks of study initiation
* History of enhanced bleeding tendency
* History of heparin-induced thrombocytopenia
* History of serious drug-related reactions, including hypersensitivity

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To determine whether direct intrapulmonary delivery of rhAPC can inhibit LPS-induced lung inflammation, thereby avoiding systemic APC effects | 1 year

SECONDARY OUTCOMES:
1. Neutrophil responses 2. Response of alveolar macrophages 3. Activation of the cytokine and chemokine network 4. Activation of coagulation and fibrinolysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tom Van der Poll, MD PhD, Principal Investigator — AMC/UvA Amsterdam
Locations (1):
- Academic Medical Center/ University of Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Kager LM, de Boer JD, Bresser P, van der Zee JS, Zeerleder S, Meijers JC, van 't Veer C, van der Poll T. Intrabronchial activated protein C enhances lipopolysaccharide-induced pulmonary responses. Eur Respir J. 2013 Jul;42(1):188-97. doi: 10.1183/09031936.00057112. Epub 2012 Oct 11. PMID 23060625